CLINICAL TRIAL: NCT01217398
Title: Phase II Single-Center Study of Bevacizumab in Combination With Temozolomide in Patients With First-Line Metastatic Uveal Melanoma
Brief Title: Temozolomide and Bevacizumab in Treating Patients With Metastatic Melanoma of the Eye
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000683852; CLCC-IC-2009-01; EUDRACT-2009-011751-46; EU-21063
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2012-08

CONDITIONS: Intraocular Melanoma
Keywords: ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size; iris melanoma; metastatic intraocular melanoma; stage IV intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Bevacizumab; Temozolomide; Amplified Fragment Length Polymorphism Analysis; Pharmacogenomic Testing

INTERVENTIONS:
Biological: bevacizumab
Drug: temozolomide
Genetic: polymorphism analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving temozolomide together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying giving temozolomide together with bevacizumab to see how well they work in treating patients with metastatic melanoma of the eye.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of temozolomide in combination with bevacizumab in treating patients with metastatic uveal melanoma not amenable to curative surgery.

Secondary

* To determine response rate in these patients.
* To determine duration of response in these patients.
* To determine progression-free survival of these patients.
* To determine overall survival of these patients.
* To determine the safety of treatment with this regimen in these patients.
* To study the CT perfusion imaging for functional imaging of response in these patients.
* To determine the pharmacogenetic influence of constitutional VEGF-A polymorphism on the efficacy and toxicity of bevacizumab. (ancillary)

OUTLINE: Patients receive oral temozolomide once daily on days 1-7 and 15-21 and bevacizumab IV over 30-90 minutes on days 8 and 22. Treatment repeats every 28 days for up to 6 courses. Patients achieving at least stable disease then receive bevacizumab monotherapy IV every 2 weeks as maintenance therapy in the absence of unacceptable toxicity and disease progression. Patients undergo CT perfusion imaging at baseline, day 28, and at 3 and 6 months.

Blood samples are collected at baseline and then periodically for VEGF-A genetic polymorphism analysis.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed uveal melanoma

  * Metastatic disease
* Measurable disease, defined as ≥ 1 measurable lesion as measured by RECIST criteria
* No curative surgical treatment envisaged
* No active brain metastases (if clinical suspicion, must have a brain CT scan within 28 days)

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR calculated creatinine clearance ≥ 50 mL/min
* Proteinuria < 2+ on urinary dipstick OR 24-hour proteinuria ≤ 1 g
* Total bilirubin ≤ 1.5 times ULN
* AST/ALT ≤ 2.5 times ULN
* Lactate dehydrogenase ≤ 5 times ULN
* INR and PT ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No uncontrolled active disease or at risk of bleeding, ongoing infection, or clotting disorder
* No other cancer except for skin carcinomas and cervical carcinoma in situ
* No pre-existing peripheral neuropathy, > grade 2 (NCI CTC-AE)
* No failure to comply with the medical follow-up of the study for geographical, social, or psychological reasons
* No recent thrombophlebitis or pulmonary embolism within the past 6 months
* No uncontrolled hypertension (systolic BP > 150 mm Hg and/or diastolic BP > 100 mm Hg)
* No concurrent active cardiovascular disease, uncontrolled by medical treatment within the past 6 months, including any of the following:

  * Unstable angina
  * Severe hypertension
  * Severe arrhythmia
* No unhealed wound, active peptic ulcer, bone fracture, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No known hypersensitivity to bevacizumab, temozolomide, or their excipients

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease
* At least 24 hours since insertion of central infusion port
* More than 5 days since prior non-hepatic biopsy or aspiration cytology
* More than 10 days since prior aspirin (> 325 mg/day), clopidogrel (> 75 mg/day), or full-dose oral or parenteral anticoagulant therapy, except prophylactic anticoagulant therapy prior to inclusion in the study
* More than 14 days since prior laparoscopic liver biopsy
* More than 28 days since prior major surgery
* More than 28 days since prior participation in another study with experimental treatment
* No other concurrent anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Disease control rate, in terms of objective response rate and the stable disease rate determined according to RECIST criteria at 6 months

SECONDARY OUTCOMES:
Response rate
Duration of response
Progression-free survival
Overall survival
Safety of this regimen in these patients
Functional imaging of response by CT perfusion imaging

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Piperno-Neumann, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France